CLINICAL TRIAL: NCT02459704
Title: Semilunar Coronally Positioned Flap With or Without Enamel Matrix Derivative for the Treatment of Miller Class I Gingival Recessions: Randomized Clinical Trial
Brief Title: Semilunar Coronally Positioned Flap With or Without Enamel Matrix Derivative for the Treatment of Gingival Recessions
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Campinas, Brazil (Other)
Responsible Party: Principal Investigator, Enilson Antonio Sallum, Professor, department of Periodontics, Piracicaba Dental School, State University of Campinas (UNICAMP), Piracicaba, São Paulo, Brazil, University of Campinas, Brazil
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 038/2012; 2013/13098-9 (Other Grant/Funding Number: FAPESP)
Record Dates: First submitted 2015-05-25; First posted 2015-06-02 (Estimated); Last update posted 2015-10-08 (Estimated); Status verified 2015-05

CONDITIONS: Gingival Recession
Keywords: Gingival Recession; Semilunar flap; Enamel matrix derivative; Periodontal regeneration
MeSH Terms: conditions — Gingival Recession

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- SCPF + EMD (TEST) (Experimental): Semilunar coronally positioned flap with Enamel matrix derivative (Emdogain)
  Interventions: Procedure: Semilunar coronally positioned flap; Device: Enamel matrix derivative (Emdogain)
- SCPF (CONTROL) (Active Comparator): Semilunar coronally positioned flap alone
  Interventions: Procedure: Semilunar coronally positioned flap

INTERVENTIONS:
Procedure: Semilunar coronally positioned flap — Semilunar coronally positioned flap with enamel matrix derivative (Emdogain) or alone.
Device: Enamel matrix derivative (Emdogain) — Enamel matrix derivative associated to semilunar coronally positioned flap (SCPF + EMD - test group)
  Arms: SCPF + EMD (TEST)

SUMMARY:
The aim of this study will be evaluate clinically the use of the Semilunar Coronally Positioned Flap (SCPF) for the treatment of gingival recessions, with or without Enamel Matrix Derivative (EMD). Thirty patients will be assigned in two groups. Half of patients will receive EMD associated to SCPF, while the other half, will receive SCPF alone.

DETAILED DESCRIPTION:
The aim of this study will be evaluate clinically the use of the Semilunar Coronally Positioned Flap (SCPF) for the treatment of gingival recessions, with or without Enamel Matrix Derivative (EMD). Thirty patients will be selected, randomized and allocated in two groups: test group (SCPF + EMD) and control group (SCPF). The subjects will should present buccal Miller class I gingival recessions with height greater than or equal to 2.0 mm and less than to 4.0 mm in maxillary canines or premolars. Clinical parameters will be evaluated: gingival recession height (GRH), gingival recession width(GRW), clinical attachment level (CAL), probing depth (PD), height (HKT) and thickness (TKT) of keratinized tissue and papillas height (HP) and width(LP), as well as plaque and gingival index. These data will be collected at baseline and 180 days after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years;
* Presence of at least one Miller Class I gingival recession ≥ 2 mm or ≤ 4mm in maxillary canines or premolars with identifiable cementum-enamel junction (CEJ);
* Height of keratinized tissue ≥ 2 mm;
* Aesthetic complaint and/or presence of dentin hypersensitivity to air stimulus;
* Full-mouth visible plaque index ≤ 20% (Ainamo & Bay 1975);
* Full-mouth sulcus bleeding index ≤ 20% (Mühlemann & Son 1971).

Exclusion Criteria:

* Smoking;
* Pregnancy;
* Presence of systemic disorders (diabetes, hypertension, heart disease or any other condition that could contraindicate periodontal surgery);
* Use of medications (immunosuppressants, phenytoin or anything else that might affect mucosal healing and repair);
* Previous periodontal surgery in the area.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2014-06; Primary Completion 2015-06 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Change in Recession Reduction as measured by difference between gingival recession depth | Baseline, 12 months
  Measured as a difference between gingival recession depth at baseline and gingival recession at 6 months follow-up.

SECONDARY OUTCOMES:
Complete root coverage | 12 months
  Assessed as percentage of sites with complete root coverage

CONTACTS AND LOCATIONS:
Overall Officials: Enilson A Sallum, PhD, Principal Investigator — University of Campinas, Brazil
Locations (1):
- Piracicaba Dental School, State University of Campinas, Piracicaba, São Paulo, Brazil

REFERENCES:
- [Derived] Franca-Grohmann IL, Sangiorgio JPM, Bueno MR, Casarin RCV, Silverio KG, Nociti FH Jr, Casati MZ, Sallum EA. Does enamel matrix derivative application improve clinical outcomes after semilunar flap surgery? A randomized clinical trial. Clin Oral Investig. 2019 Feb;23(2):879-887. doi: 10.1007/s00784-018-2506-y. Epub 2018 Jun 12. PMID 29948276